CLINICAL TRIAL: NCT04787263
Title: Phase I/II Study of Anti-CD19 Chimeric Antigen Receptor-Expressing T Cells in Pediatric Patients Affected by Relapsed/Refractory CD19+ Acute Lymphoblastic Leukemia and Diffuse Large B Cell Lymphoma (DLBCL) or Primary Mediastinal B Cell Lymphoma (PML)
Brief Title: CD19-CAR_Lenti T Cells in Pediatric Patients Affected by Relapsed/Refractory CD19+ ALL and DLBCL or PML
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CAR_Lenti
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma; Primary Mediastinal Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR_Lenti (Experimental): Following lymphodepletion with chemotherapy (fludarabine + cyclophosphamide), patients will be treated with 1.0 to 3.0 x 10^6/kg CD19-Chimeric Antigen Receptor (CAR)_Lenti positive cells as a single dose. The product will be infused fresh, at the end of manufacturing.
  Interventions: Biological: CD19-CAR_Lenti T cell

INTERVENTIONS:
Biological: CD19-CAR_Lenti T cell — Fresh peripheral blood mononuclear cells are manufactured to obtain CD19-CAR_Lenti T cell, second generation CAR T cells incorporating the 4-1BB costimulatory domain. The fresh product is infused following lymphodepletion chemotherapy at a dose of 1.0-3.0x10^6 CAR+ cells/kg.

SUMMARY:
This study aims at evaluating the feasibility and safety of the administration of autologous T cells that have been modified through the introduction of a chimeric antigen receptor targeting the B-cell surface antigen CD19, following administration of lymphodepleting chemotherapy regimen, in children and adults with relapsed/refractory B-cell acute lymphoblastic leukemia (B- ALL) or aggressive B-cell Non-Hodgkin lymphoma (B-NHL). The phase II extension is aimed at testing the efficacy of the treatment at the optimal dose defined in the phase I. In addition, the investigators hypothesize that it is feasible to successfully manufacture CAR T cells to meet the established release criteria at a maximum target dose of 3.0 x 10^6 cells/kilogram recipient total body weight in this patient population using the Miltenyi CliniMACS Prodigy® closed transduction system.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD19 expressing B-ALL or DLBCL or PML and one of the following:

   1. Patients in 1st relapse, with High-Risk (HR) features including: MLL- rearrangements, E2A/TCF3-PBX1, TCF3-HLF [t(17;19)], hypodiploidy (i.e., <44 chromosomes), TP53 alterations, early (i.e., <30 months from diagnosis)/very early (i.e., <18 months from diagnosis) isolated or combined bone marrow relapse
   2. MRD > 0.1% after either reinduction therapy or any course of consolidation for relapsed ALL
   3. Patients with DLBCL or PML in 1st or subsequent relapse, after at least one standard frontline chemotherapy
2. Age: 1 year - 25 years for Bcp-ALL and 1-35 years for B-NHL.
3. Voluntary informed consent is given. For subjects < 18 year-old their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
4. Clinical performance status: Patients > 16 years of age: Karnofsky greater than or equal to 60%; Patients < 16 years of age: Lansky scale greater than or equal to 60%.
5. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
6. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe, uncontrolled active infections
3. HIV, or active HCV and/or HBV infection (detection of viral RNA/DNA in blood)
4. Life-expectancy < 6 weeks
5. Hepatic function: Inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6 x ULN
6. Renal function: serum creatinine > 3x ULN for age.
7. Blood oxygen saturation < 90%.
8. Cardiac function: Left ventricular ejection fraction lower than 45% by ECHO.
9. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject.
10. BM blasts > 50% pre-infusion.
11. Hyperleukocytosis (greater than or equal to 20,000 blasts/microliter) or rapidly progressive disease that in the evaluation of the investigator would compromise ability to complete study therapy
12. Presence of active, grade 2-4 acute or moderate-severe chronic GvHD
13. Recurrent or refractory ALL with testicular involvement
14. Concurrent or recent prior therapies, before infusion:

    1. Systemic steroids (at a dose > 2 mg/kg prednisone) in the 2 weeks before infusion. Recent or current use of inhaled/topical/non-absorbable steroids is not exclusionary.
    2. Systemic chemotherapy in the week preceding infusion.
    3. Anti-thymocyte globulin (ATG) in the 4 weeks preceding infusion.
    4. Immunosuppressive agents in the 1 week preceding infusion.
    5. Radiation therapy must have been completed at least 3 weeks prior to enrollment.
    6. Other anti-neoplastic investigational agents currently administered or within 30 days prior to infusion (i.e. start of protocol therapy);
    7. Exceptions:

    i. There is no time restriction with respect to prior intrathecal chemotherapy, provided that there is complete recovery from any acute toxic effects of such; ii. Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study provided that they meet all other eligibility criteria; iii. Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided that there has been no increase in dose for at least 2 weeks prior to starting apheresis;
15. Patient-derived CD19-CAR_Lenti production failure: vitality of the fresh product <80%, CD3+ cells <80%, CD3+ CAR+ cells <10%, non-sterility in IPC at day 5, endotoxin contamination (> 5 EU/ml) in IPC at day 5, mycoplasma contamination in IPC at day 5, failure of the visual inspection.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2038-03-03 (Estimated)

PRIMARY OUTCOMES:
Phase I - Identification of dose limiting toxicities (DLTs) and recommended dose (RD) | 4 weeks after CAR T cell infusion
  Toxicity will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 5.0
Phase I - Identification of recommended dose (RD) | 4 weeks after CAR T cell infusion of the last patient in the last dose level
  The recommended dose of CD19-CAR_Lenti will be defined as the maximum tolerated dose (MTD) or the highest dose studied, if an MTD is not reached.
Phase II - Efficacy | Up to 6 months after CAR T cell infusion
  Bone marrow morphological and minimal residual disease complete remission rate at day 28 after infusion for BCP-ALL; Overall Response Rate (CR, CRi, PR and SD) at day 28, day 90 and day 180 after CAR T cells infusion

SECONDARY OUTCOMES:
Relapse Rate (RR) | Up to 2 years
Overall survival (OS) | Up to 2 years
Disease-Free Survival (DFS) | Up to 2 years
In vivo persistence/expansion of infused CAR T cell | Up to 2 years
  Detection of infused CAR T cell in the peripheral and bone marrow blood
Cytokine profiling | Up to 10 days after CAR T cell infusion
  Define serum cytokine profile (Th1/Th2) after T cell infusion and correlation with cytokine release syndrome (CRS)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Pediatrico Bambino Gesù, Roma, Italy